CLINICAL TRIAL: NCT02968758
Title: Prospective Multi-Center Study for Clinical Validation of the Molecular-Based GenePOC CDiff System for the Detection of Toxin B Gene From Toxigenic Clostridium Difficile Strains in Unformed (Soft or Liquid) Human Stool Specimens
Brief Title: Validation of the GenePOC CDiff Assay for the Detection of the Toxin B Gene From Toxigenic Clostridium Difficile Strains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GenePOC CDiff_clinical-01
Record Dates: First submitted 2016-11-15; First posted 2016-11-21 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2019-01

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Accuracy Testing (Experimental): Comparison between GenePOC PCR and Reference Method
  Interventions: Device: Comparison between GenePOC PCR and Reference Method

INTERVENTIONS:
Device: Comparison between GenePOC PCR and Reference Method — Stool specimen will be tested with the GenePOC CDiff test on the GenePOC Instrument. The results will be compared to Reference Method defined as direct and enriched culture method for observation of a toxigenic Clostridium difficile strain.

SUMMARY:
The primary purpose of this clinical investigation is to verify the performance of the GenePOC CDiff test on the GenePOC instrument. This will be achieved by comparing the GenePOC CDiff test to the Toxigenic Culture (TC) and cell cytotoxicity neutralisation assay (CCNA), a conventional method considered as gold standard for detection of toxigenic Clostridium difficile in stool specimens.

DETAILED DESCRIPTION:
The GenePOC CDiff test performed on the GenePOC™ instrument is a qualitative in vitro diagnostic (IVD) test that utilizes automated sample preparation and real-time polymerase chain reaction (rtPCR) to detect the toxin B (tcdB) gene of toxigenic Clostridium difficile (C. difficile) in unformed (liquid or soft) stool specimens obtained from patients suspected of having C. difficile infection (CDI).

The GenePOC CDiff system comprises the GenePOC instrument and the GenePOC CDiff test, which consists of:

1. Transfer Loop (TL)
2. CDiff disposable microfluidic cartridges (PIE) (described in this document as PIEs because of the shape of the cartridge)
3. CDiff Sample Buffer Tube (SBT)
4. Disposable Transfer Tool (DTT).

The GenePOC Instrument is fully automated and integrates sample lysis, dilution, amplification and detection of the target sequence in complex samples using real-time Polymerase chain reaction (rtPCR). User intervention is only required for discharging the patient sample into the SBT (sample Buffer Tube), transferring the sample into the PIE and for loading/unloading the PIEs into the instrument. The GenePOC instrument consists of a rotor to spin the PIEs, temperature control, fluorescence detection, a tactile user-friendly interface, two barcode readers, and integrated firmware and software to deliver results to the user. The PIE is a closed system that prevents the risk of contamination.

An unformed (soft or liquid) stool specimen is collected using standard stool collection device. Using a disposable 5µL inoculating loop (transfer loop) dipped into the homogenized stool specimen, stool material is transferred into SBT and vortexed. Sample is then transferred to the GenePOC CDiff PIE. The GenePOC CDiff PIE is then automatically processed by the GenePOC Instrument. On completion of a run, the user removes the processed PIEs from the instrument and discards them according to local biological waste management procedures.

One GenePOC instrument per site will be allocated. The purpose of the clinical investigation is to enroll sufficient specimens from up to 7 Clinical Centers to obtain a total of 150 specimens positive for CDiff based on the Reference Method final result.

Subject Informed consent is not required for this clinical trial as the testing will be performed on excess de-identified specimens only.

ELIGIBILITY:
Inclusion Criteria:

* Unformed Stool specimens from patients suspected of having CDI for whom diagnostic tests are indicated and ordered;
* At least 1.25mL of unformed stool specimen (defined as specimen assuming the shape of its container);
* Only one (1) specimen per patient will be included in the study;
* Materials use within their expiration date;
* Transport, storage times, and conditions (e.g. room temperature and/or refrigerated) within requested indications.

Exclusion Criteria:

* Specimens from patients for whom CDI diagnostic tests have not been ordered;
* Transport and storage times and conditions that exceed these Study Protocol requirements;
* Formed or hard stool specimens or rectal swabs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2461 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Allibert, Study Director — Meridian Bioscience, Inc.
Locations (7):
- United States (5):
  - Wishard Health Services, Indianapolis, Indiana
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Detroit Medical Center University Laboratories, Detroit, Michigan
  - Tricore Laboratory University of New Mexico, Albuquerque, New Mexico
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Mount Sinai Hospital Joseph and Wolf Lebovic Health Complex, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Accuracy Testing - Fresh Specimen: Comparison between GenePOC PCR and Reference Method
  Comparison between GenePOC PCR and Reference Method: Fresh Stool specimen will be tested with the GenePOC CDiff test on the GenePOC Instrument. The results will be compared to Reference Method defined as direct and enriched culture method for observation of a toxigenic Clostridium difficile strain.
- Accuracy Testing - Frozen Specimen: Comparison between GenePOC PCR and Reference Method
  Comparison between GenePOC PCR and Reference Method: Frozen Stool specimen will be tested with the GenePOC CDiff test on the GenePOC Instrument. The results will be compared to Reference Method defined as direct and enriched culture method for observation of a toxigenic Clostridium difficile strain.
Period: Overall Study
Arm/Group | Accuracy Testing - Fresh Specimen | Accuracy Testing - Frozen Specimen
Started | 797 | 1664
Completed | 797 | 1664
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all specimens were included
Groups:
- Total: Total of all reporting groups
Arm/Group | Accuracy Testing - Fresh Specimen | Accuracy Testing - Frozen Specimen | Total
Number analyzed (Participants) | 797 | 1664 | 2461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 80 | 114
  Between 18 and 65 years | 399 | 800 | 1199
  >=65 years | 364 | 784 | 1148
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Gender information was not collected during the trial.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 79 | 0 | 79
  United States | 718 | 1664 | 2382

OUTCOME MEASURES:

1. Primary Outcome: Performance Characteristics : Clinical Sensitivity (True Positive Rate) and Clinical Specificity (True Negative Rate) in Comparison to the Reference Method
Description: To establish the performance characteristics of the GenePOC CDiff System for its use in determining the presence of CDiff in liquid/unformed stool specimen obtained from patients suspected of having C. difficile infection (CDI).
  Sensitivity will be established as the proportion of positives that are correctly identified by the GenePOC CDiff System, when compared to the Reference Method.
  Specificity will be established as the proportion of negatives that are correctly identified by the GenePOC CDiff System, when compared to the Reference Method.
Time Frame: At the time of the results with Reference Method is confirmed, up to 3 months
Measure: Number (95% Confidence Interval); unit: percentage of specimens
Arm/Group | Accuracy Testing - Fresh Specimen | Accuracy Testing - Frozen Specimen
Number analyzed (Participants) | 797 | 1664
percentage of specimens
  Sensitivity | 95.5 [87.3 to 99.1] | 95.2 [90.8 to 97.9]
  Specificity | 93.4 [91.4 to 95.1] | 95.3 [94.1 to 96.3]

2. Secondary Outcome: Positive and Negative Predictive Values (PPV and NPV)
Description: To estimate the Positive and Negative Predictive Values (PPV and NPV) of the GenePOC CDiff System.
  PPV is the percentage of true positives out of all positive results (true positive/true positive + false positive).
  NPV is the percentage of true negatives out of all negative results (true negative/true negative +false negative.).
Time Frame: At the time of the results with Reference Method is confirmed, up to 3 months
Measure: Number (95% Confidence Interval); unit: percentage of specimens
Arm/Group | Accuracy Testing - Fresh Specimen | Accuracy Testing - Frozen Specimen
Number analyzed (Participants) | 797 | 1664
percentage of specimens
  PPV | 82.0 [73.6 to 88.6] | 83.1 [77.7 to 87.7]
  NPV | 96.8 [95.2 to 98.0] | 98.0 [97.2 to 98.7]

3. Secondary Outcome: Unresolved Sample Results
Description: To estimate the rate of unresolved results for the GenePOC CDiff System due to Sample Processing control failure (unresolved sample results).
Time Frame: At the time of the results with Reference Method is confirmed, up to 3 months
Measure: Number (95% Confidence Interval); unit: percentage of Unresolved
Arm/Group | Accuracy Testing - Fresh Specimen | Accuracy Testing - Frozen Specimen
Number analyzed (Participants) | 797 | 1664
percentage of Unresolved | 1.1 [0.52 to 2.13] | 0.8 [0.42 to 1.33]

4. Secondary Outcome: Indeterminate Sample Results
Description: To estimate the rate of indeterminate results for the GenePOC CDiff Test due to an Instrument failure (indeterminate sample results).
Time Frame: At the time of the results with Reference Method is confirmed, up to 3 months
Measure: Number (95% Confidence Interval); unit: percentage of Indeterminates
Arm/Group | Accuracy Testing - Fresh Specimen | Accuracy Testing - Frozen Specimen
Number analyzed (Participants) | 797 | 1664
percentage of Indeterminates | 1.6 [1.16 to 2.20] | 1.5 [0.78 to 2.61]

ADVERSE EVENTS:
Time Frame: Adverse event were assessed at the time of individual patient enrollment and participation, which lasts approximately 1-2 minutes at most.
Description: Adverse event procedures were established at each site, but no adverse event was observed nor reported during the enrollment period.
Arm/Group | Accuracy Testing
All-Cause Mortality (participants affected / at risk) | 0/2461
Serious Adverse Events (participants affected / at risk) | 0/2461
Other Adverse Events (participants affected / at risk) | 0/2461

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02968758/Prot_SAP_000.pdf